CLINICAL TRIAL: NCT06541743
Title: Efficacy of Regular, Musical and Electric Toothbrushes in Plaque Removal in Children - A Randomized Clinical Trial
Brief Title: Efficacy of Regular, Musical and Electric Toothbrushes in Plaque Removal in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jouf University (Other)
Responsible Party: Principal Investigator, Rakhi Issrani, lecturer, Jouf University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: (DGSSR-2023-01-02524)
Record Dates: First submitted 2024-07-17; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Children, Adult; Plaque
Keywords: Children; Oral Health; Toothbrush; Plaque Removal
MeSH Terms: conditions — Plaque, Amyloid

STUDY DESIGN:
Intervention Model Description: * (Regular Toothbrush): Oral-B Chhota Bheem Toothbrush.
  * (Musical Toothbrush): Aqua White Musical Chhota Bheem Toothbrush.
  * (Electric Toothbrush): Oral-B Star Wars Kids Electric Toothbrush
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Regular Toothbrush (Active Comparator): Oral-B Chhota Bheem Toothbrush.
  Interventions: Device: Regular Toothbrush
- Musical Toothbrush (Active Comparator): Aqua White Musical Chhota Bheem Toothbrush.
  Interventions: Device: Musical toothbrush
- Electric Toothbrush (Active Comparator): Oral-B Star Wars Kids Electric Toothbrush.
  Interventions: Device: Electric toothbrush

INTERVENTIONS:
Device: Regular Toothbrush — Participants and their guardians will be instructed in the horizontal scrub technique and asked to adhere to a brushing regimen of two minutes, twice daily, for 45 days. Standard fluoride toothpaste and a diary for recording brushing experiences will also provided. Guardians will be supervised brushing to ensure compliance and prevent the use of other oral hygiene measures.
  Arms: Regular Toothbrush
Device: Musical toothbrush — Participants and their guardians will be instructed in the horizontal scrub technique and asked to adhere to a brushing regimen of two minutes, twice daily, for 45 days. Standard fluoride toothpaste and a diary for recording brushing experiences will also provided. Guardians will be supervised brushing to ensure compliance and prevent the use of other oral hygiene measures.
  Arms: Musical Toothbrush
Device: Electric toothbrush — Participants and their guardians will be instructed in the horizontal scrub technique and asked to adhere to a brushing regimen of two minutes, twice daily, for 45 days. Standard fluoride toothpaste and a diary for recording brushing experiences will also provided. Guardians will be supervised brushing to ensure compliance and prevent the use of other oral hygiene measures.
  Arms: Electric Toothbrush

SUMMARY:
Tooth brushing is essential for maintaining oral hygiene, especially in children, who are at a critical stage for developing lifelong oral health habits. Establishing effective tooth brushing behaviors for school-aged children (6-12 years) is vital for long-term dental health. Consistent and effective tooth brushing is crucial for reducing supragingival plaque, which is key to preventing periodontal diseases and ensuring good oral hygiene. Despite the availability of various plaque control methods, tooth brushing remains the most effective and safest approach.

However, young children, particularly those under ten, often struggle with the dexterity and motivation needed for proper tooth brushing, resulting in inadequate plaque removal. Manual tooth brushing, though effective, can become monotonous and fail to engage children, making it difficult to establish regular brushing habits. Studies have shown that regular removal of supragingival plaque can significantly reduce both supra- and subgingival pathogenic species, underscoring the importance of effective plaque control.

Innovative solutions such as electric and musical toothbrushes have been developed to address these challenges.

DETAILED DESCRIPTION:
Electric toothbrushes enhance plaque removal through mechanical action, while musical toothbrushes aim to boost motivation and compliance by incorporating interactive elements like music and colorful designs. Musical toothbrushes play music for two minutes, encouraging children to brush for the recommended duration and making the activity more enjoyable. Previous research has shown varying levels of success with these advanced toothbrushes. For example, one of the recent study have found that musical toothbrushes significantly improved plaque control compared to regular ones. Similarly, other studies have reported substantial plaque reduction with musical toothbrushes. Furthermore, it has been observed that while both manual and powered toothbrushes improved clinical parameters, powered toothbrushes had a more significant impact on gingival health.

Despite these promising results, there is a lack of comprehensive comparative studies on the efficacy of regular, electric, and musical toothbrushes in children. This study aimed to address this gap by conducting a randomized clinical trial to evaluate and compare the effectiveness of these three types of toothbrushes in removing supragingival plaque in children aged 6-12 years.

To the best of our knowledge, this is the first clinical study wherein the comparisons had been made between regular, musical and electric toothbrushes. The findings will provide valuable insights into the most effective tools for promoting oral hygiene in children, potentially shaping future recommendations and practices in pediatric dentistry.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-12 years;
* Cooperative children; and
* Children with a minimum of twenty teeth

Exclusion Criteria:

* Children with poor oral hygiene characterized by extrinsic stains or calculus deposits;
* Presence of any oral lesions;
* Presence of malocclusion; and
* Medically compromised patients

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 111 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Plaque Index (Quigley and Hein) | 45 days
  Plaque assessments was conducted at baseline (day 0) and on days 15, 30, and 45. Participants were refrain from oral hygiene for 24 hours before each recall visit. During each visit, they were supposed to brush under supervision for two minutes with their assigned toothbrush and toothpaste. Plaque disclosure was achieved using a 5 mL disclosing solution for 15 seconds, followed by rinsing with 10 mL water for 10 seconds.
  Quigley-Hain plaque index
  0
  No plaque
  1
  Isolated flecks of plaque at the gingival margin
  2
  A continuous band of plaque up to 1mm at the gingival margin
  3
  Plaque greater than 1mm in width and covering up to one third of the tooth surface
  4
  Plaque covering from one thirds to two thirds of the tooth surface
  5
  Plaque covering more than two thirds of the tooth surface

CONTACTS AND LOCATIONS:
Overall Officials: Namdeo Prabhu, MDS, Study Chair — College of Dentistry, Jouf University
Locations (1):
- College of Dentistry, Jouf University, Sakakah, Al Jawf Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kitsaras G, Goodwin M, Kelly MP, Pretty IA. Bedtime Oral Hygiene Behaviours, Dietary Habits and Children's Dental Health. Children (Basel). 2021 May 19;8(5):416. doi: 10.3390/children8050416. PMID 34069504
- [Background] Axe A, Mueller WD, Rafferty H, Lang T, Gaengler P. Impact of manual toothbrush design on plaque removal efficacy. BMC Oral Health. 2023 Oct 25;23(1):796. doi: 10.1186/s12903-023-03518-6. PMID 37880662
- [Background] Feres M, Gursky LC, Faveri M, Tsuzuki CO, Figueiredo LC. Clinical and microbiological benefits of strict supragingival plaque control as part of the active phase of periodontal therapy. J Clin Periodontol. 2009 Oct;36(10):857-67. doi: 10.1111/j.1600-051X.2009.01471.x. Epub 2009 Aug 23. PMID 19703236
- [Background] Mateu FA, Boneta AE, DeVizio W, Stewart B, Proskin HM. A clinical investigation of the efficacy of two dentifrices for controlling established supragingival plaque and gingivitis. J Clin Dent. 2008;19(3):85-94. PMID 19301514
- [Background] 5. Liu L. The impact of innovation of electric toothbrush. 2022. https://doi.org/10.2991/aebmr.k.220307.295
- [Background] Prendergast V, Chapple KM. Evaluation and Acceptance of an Electric Toothbrush Designed for Dependent Patients. Cureus. 2021 Jun 1;13(6):e15372. doi: 10.7759/cureus.15372. eCollection 2021 Jun. PMID 34249525
- [Background] Lee J, Park HM, Kim YW. Comparative Analysis of Plaque Removal and Wear between Electric-Mechanical and Bioelectric Toothbrushes. Bioengineering (Basel). 2024 May 9;11(5):474. doi: 10.3390/bioengineering11050474. PMID 38790341
- [Background] Vargas CM, Arevalo O. How dental care can preserve and improve oral health. Dent Clin North Am. 2009 Jul;53(3):399-420. doi: 10.1016/j.cden.2009.03.011. PMID 19482119
- [Background] Ganesh M, Shah S, Parikh D, Choudhary P, Bhaskar V. The effectiveness of a musical toothbrush for dental plaque removal: a comparative study. J Indian Soc Pedod Prev Dent. 2012 Apr-Jun;30(2):139-45. doi: 10.4103/0970-4388.99988. PMID 22918099
- [Background] 10. Pillay R, Mathur A, Jain M, Singh A, Gupta V. Comparative efficacy of musical and regular toothbrush in children. Int J Curr Res Rev. 2021;13(14):142-7.
- [Background] Subburaman N, Madan Kumar PD, Iyer K. Effectiveness of musical toothbrush on oral debris and gingival bleeding among 6-10-year-old children: A randomized controlled trial. Indian J Dent Res. 2019 Mar-Apr;30(2):196-199. doi: 10.4103/ijdr.IJDR_128_17. PMID 31169149
- [Background] Haffajee AD, Thompson M, Torresyap G, Guerrero D, Socransky SS. Efficacy of manual and powered toothbrushes (I). Effect on clinical parameters. J Clin Periodontol. 2001 Oct;28(10):937-46. doi: 10.1034/j.1600-051x.2001.028010937.x. PMID 11686812

DOCUMENTS (1):
  • Study Protocol (2024-08-03): https://cdn.clinicaltrials.gov/large-docs/43/NCT06541743/Prot_000.pdf